CLINICAL TRIAL: NCT04588428
Title: Study to Evaluate the Safety, Tolerability and Immunogenicity of INO-4700 for Middle East Respiratory Syndrome Coronavirus (MERS-CoV) in Healthy Volunteers
Brief Title: Safety, Tolerability and Immunogenicity of INO-4700 for MERS-CoV in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MERS-201
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Middle East Respiratory Syndrome Coronavirus (MERS-CoV)
Keywords: Healthy; Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (10):
- Part 1: INO-4700 Group A (Experimental): Participants received one intradermal (ID) injection of 0.6 milligram (mg) of INO-4700 followed by electroporation (EP) using the CELLECTRA™ 2000 device on Day 0 and Week 4.
  Interventions: Drug: INO-4700; Device: CELLECTRA™ 2000
- Part 1: INO-4700 Group B (Experimental): Participants received one ID injection of 1.0 mg of INO-4700 followed by EP using the CELLECTRA™ 2000 device on Day 0 and Week 4.
  Interventions: Drug: INO-4700; Device: CELLECTRA™ 2000
- Part 1: INO-4700 Group C (Experimental): Participants received one ID injection of 1.0 mg of INO-4700 followed by EP using the CELLECTRA™ 2000 device on Day 0 and Week 8.
  Interventions: Drug: INO-4700; Device: CELLECTRA™ 2000
- Part 1: INO-4700 Group D (Experimental): Participants received two ID injections (in an acceptable location on two different limbs) of 0.5 mg each of INO-4700 followed by EP using the CELLECTRA™ 2000 device on Day 0 and Week 8.
  Interventions: Drug: INO-4700; Device: CELLECTRA™ 2000
- Part 1: INO-4700 Group E (Experimental): Participants received two ID injections (in an acceptable location on two different limbs) of 1.0 mg each of INO-4700 followed by EP using the CELLECTRA™ 2000 device on Day 0 and Week 4.
  Interventions: Drug: INO-4700; Device: CELLECTRA™ 2000
- Part 1: Placebo Group F (Placebo Comparator): Participants received one ID injection of placebo followed by EP using the CELLECTRA™ 2000 device on Day 0 and Week 4.
  Interventions: Drug: Placebo; Device: CELLECTRA™ 2000
- Part 1: Placebo Group G (Placebo Comparator): Participants received one ID injection of placebo followed by EP using the CELLECTRA™ 2000 device on Day 0 and Week 8.
  Interventions: Drug: Placebo; Device: CELLECTRA™ 2000
- Part 1: Placebo Group H (Placebo Comparator): Participants received two ID injections (in an acceptable location on two different limbs) of placebo followed by EP using the CELLECTRA™ 2000 device on Day 0 and Week 8.
  Interventions: Drug: Placebo; Device: CELLECTRA™ 2000
- Part 1: Placebo Group I (Placebo Comparator): Participants received two ID injections (in an acceptable location on two different limbs) of placebo followed by EP using the CELLECTRA™ 2000 device on Day 0 and Week 4.
  Interventions: Drug: Placebo; Device: CELLECTRA™ 2000
- Part 2: Parts 2A and 2B (Experimental): Participants were planned to receive ID injection of INO-4700 based on optimal dose and regimen selection in Part 1 followed by EP using the CELLECTRA™ 2000 device on Day 0, Week 4 or Week 8 and a booster dose at Week 48 (only for Part 2B participants were planned to receive a third dose).
  Interventions: Drug: INO-4700; Device: CELLECTRA™ 2000

INTERVENTIONS:
Drug: INO-4700 — INO-4700 was administered ID.
  Arms: Part 1: INO-4700 Group A; Part 1: INO-4700 Group B; Part 1: INO-4700 Group C; Part 1: INO-4700 Group D; Part 1: INO-4700 Group E
Drug: Placebo — Sterile saline sodium citrate (SSC) buffer (SSC-0001) was administered ID.
  Other Names: SSC-0001
  Arms: Part 1: Placebo Group F; Part 1: Placebo Group G; Part 1: Placebo Group H; Part 1: Placebo Group I
Device: CELLECTRA™ 2000 — EP using the CELLECTRA™ 2000 device was administered following ID drug administration
  Arms: Part 1: INO-4700 Group A; Part 1: INO-4700 Group B; Part 1: INO-4700 Group C; Part 1: INO-4700 Group D; Part 1: INO-4700 Group E; Part 1: Placebo Group F; Part 1: Placebo Group G; Part 1: Placebo Group H; Part 1: Placebo Group I
Drug: INO-4700 — INO-4700
  Arms: Part 2: Parts 2A and 2B
Device: CELLECTRA™ 2000 — CELLECTRA™ 2000
  Arms: Part 2: Parts 2A and 2B

SUMMARY:
The purpose of this Phase 2a, randomized, blinded, placebo-controlled, multi-center study is to evaluate the safety, tolerability and immunogenicity of INO-4700 administered by intradermal (ID) injection followed by electroporation (EP) using the CELLECTRA™ 2000 device in healthy adult volunteers for Middle East Respiratory Syndrome Coronavirus (MERS-CoV) infection. This study was divided into 2 parts: Part 1- dose finding stage and Part 2- dose expansion stage.

ELIGIBILITY:
Key Inclusion Criteria:

* Judged to be healthy by the Investigator on the basis of medical history, physical examination and vital signs performed at Screening;
* Able and willing to comply with all study procedures;
* Screening laboratory results within normal limits;
* Negative tests for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody and Human Immunodeficiency Virus (HIV) antibody;
* Screening electrocardiogram (ECG) deemed by the Investigator as having no clinically significant findings (e.g. Wolff-Parkinson-White syndrome);
* Be post-menopausal or be surgically sterile or have a partner who is sterile or use medically effective contraception with a failure rate of < 1% per year when used consistently and correctly from screening until 3 months following last dose.

Key Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant or father children within the projected duration of the trial starting with the screening visit until 3 months following last dose;
* History of respiratory diseases such as asthma, chronic obstructive pulmonary disease (COPD) or chronic bronchitis;
* Currently participating in or has participated in a study with an investigational product within 30 days preceding Day 0;
* Previous receipt of any vaccine within 30 days preceding Day 0 or planning to receive any vaccine during the timeframe restricted per the protocol;
* Previous receipt of an investigational vaccine product for the prevention of MERS;
* Prior exposure to MERS-CoV or camels;
* Participants who participate in MERS-201 Part 1 cannot participate in MERS-201 Part 2;
* Fewer than two acceptable sites available for ID injection and EP considering the deltoid and anterolateral quadriceps muscles;
* Prisoner or participants who are compulsorily detained (involuntary incarceration);
* Current or anticipated concomitant immunosuppressive therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids) prior to dosing. Systemic corticosteroids must be discontinued at least 3 months prior to first dose;
* Reported active drug or alcohol or substance abuse or dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventure Orizu, MD, Study Director — Inovio Pharmaceuticals
Locations (6):
- Jordan (2):
  - Clinical Research Center, Irbid Specialty Hospital (CRC/ISH), Irbid
  - Pharmaceutical Research Center / Jordan University of Science and Technology, Irbid
- Kenya (2):
  - Kenya Medical Research Institute (KEMRI)/Walter Reed Project (WRP), Kericho
  - Ahero Clincal Trials Unit, Kisumu
- Lebanon (2):
  - American University of Beirut Medical Center, Beirut
  - Hammoud Hospital University Medical Center, Saida

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries and all collected IPD will be stripped of identifiers and may be made available upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Anonymous IPD may be shared following or during the publication of summary data. Archival data may be accessed for up to 10 years following the end of the study.
Access Criteria: Those who request the anonymous IPD must provide a plan of study explaining how the data will be used. Requests may be sent to the Central Contact Person. Requests will be reviewed based on the potential for the planned use of the IPD for advancing scientific knowledge and theory.

REFERENCES:
- [Derived] Agnes JT, Marcus SA, Al-Ghraibeh SS, Al-Sweedan SA, Kosgei J, Ogutu B, Yang S, Walker KA, Orizu B, Broderick KE, Boyer J, Ramos S, Morrow MP, Kraynyak K, Sylvester AJ, Gillespie E, Liebowitz D, Humeau LM. Safety, tolerability, and immunogenicity of a DNA-based vaccine (INO-4700) against Middle East respiratory syndrome coronavirus: phase 2a study in healthy volunteers. Front Immunol. 2025 Nov 14;16:1662923. doi: 10.3389/fimmu.2025.1662923. eCollection 2025. PMID 41322416

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult volunteers were enrolled at 6 study sites between 21 June 2021 and 19 January 2023.
Pre-assignment Details: This study was planned for two parts i.e., Part 1 and Part 2. A total of 218 participants were screened for Part 1 of the study, out of which 192 participants were enrolled. Part 1 was to select the optimal dose for Part 2. However, none of the dose groups studied in Part 1 met the immunological criteria for advancement to Part 2. Consequently, the study ended at the conclusion of Part 1. The data is reported only for Part 1.
Period: Overall Study
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Started | 32 | 33 | 32 | 32 | 31 | 8 | 8 | 8 | 8
Completed | 32 | 33 | 29 | 31 | 31 | 7 | 8 | 8 | 8
Not Completed | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The modified intent to treat (mITT) population included all participants who received at least one dose of the INO-4700 or placebo.
Groups:
- Part 1: INO-4700 Group A: Participants received one ID injection of 0.6 mg of INO-4700 followed by EP using the CELLECTRA™ 2000 device on Day 0 and Week 4.
- Total: Total of all reporting groups
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I | Total
Number analyzed (Participants) | 32 | 33 | 32 | 32 | 31 | 8 | 8 | 8 | 8 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (7.66) | 34.2 (9.20) | 34.8 (7.69) | 31.5 (8.63) | 35.0 (7.77) | 28.4 (8.40) | 34.0 (10.62) | 30.3 (7.52) | 39.8 (6.96) | 33.8 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 11 | 10 | 16 | 0 | 4 | 3 | 2 | 68
  Male | 22 | 21 | 21 | 22 | 15 | 8 | 4 | 5 | 6 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 6 | 2 | 2 | 1 | 1 | 1 | 0 | 20
  White | 30 | 28 | 26 | 30 | 29 | 7 | 7 | 7 | 8 | 172
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs), Graded by Severity, and Treatment-related AEs
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have a causal relationship with treatment. TEAEs: AEs with onset after administration of study medication through the end of the study, or any event that was present at baseline but worsened in intensity or was subsequently considered drug-related by the Investigator through the end of the study. TEAEs were graded based on the Toxicity Grading Scale for Healthy Adult & Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (Food and Drug Administration [FDA] Guidance for Industry), as Grade 1: No interference with activity, Grade 2: Some interference with activity, Grade 3: Prevents daily activity/requires medical intervention & Grade 4: Emergency room visit/hospitalization. A causally related AE is one judged by the Investigator to have a possible, probable, or definite relationship to the administration of an investigational product (IP).
Time Frame: From the first dose of the study drug up to the end of the study (up to 48.7 weeks)
Population: The safety population included all participants who received at least one dose of INO-4700 or placebo administered by ID injection. Percentages are rounded off to the nearest decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Number analyzed (Participants) | 32 | 33 | 32 | 32 | 31 | 8 | 8 | 8 | 8
percentage of participants
  Percentage of Participants With TEAEs | 34.4 | 30.3 | 43.8 | 31.3 | 41.9 | 25.0 | 75.0 | 25.0 | 50.0
  Percentage of Participants With ≥ 1 Grade 1 TEAEs | 21.9 | 24.2 | 28.1 | 28.1 | 32.3 | 0.0 | 50.0 | 12.5 | 25.0
  Percentage of Participants With ≥ 1 Grade 2 TEAEs | 12.5 | 12.1 | 28.1 | 3.1 | 12.9 | 25.0 | 50.0 | 12.5 | 25.0
  Percentage of Participants With ≥ 1 Grade 3 TEAEs | 3.1 | 0 | 6.3 | 0.0 | 3.2 | 0.0 | 0.0 | 0.0 | 0.0
  Percentage of Participants With ≥ 1 Grade 4 TEAEs | 0.0 | 3.0 | 3.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Percentage of Participants With Treatment Related TEAEs | 3.1 | 9.1 | 0.0 | 6.3 | 3.2 | 0.0 | 0.0 | 0.0 | 12.5

2. Primary Outcome: Part 1: Percentage of Participants With Injection Site Reactions
Description: Reactions arising from the injectable product administration procedure were reported as injection site reactions. Injection site reactions were assessed in accordance with the 'Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials' FDA Guidance for Industry, September 2007. Local reactions to the injectable product such as pain, tenderness, erythema/redness, and induration/swelling were recorded. Injection site reactions were evaluated starting 30 minutes following the injection.
Time Frame: From the first dose of the study drug up to the end of the study (up to 48.7 weeks)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Number analyzed (Participants) | 32 | 33 | 32 | 32 | 31 | 8 | 8 | 8 | 8
percentage of participants
  Percentage of Participants With Injection Site Erythema | 0 | 0 | 0 | 3.1 | 0 | 0 | 0 | 0 | 0
  Percentage of Participants With Injection Site Pruritis | 0 | 3.0 | 0 | 6.3 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part 1: Percentage of Participants With Adverse Events of Special Interest (AESIs)
Description: An AESI (serious or non-serious) was defined as one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Principal Investigator to the Sponsor can be appropriate.
Time Frame: From Screening to the end of the study (up to 48.7 weeks)
Population: The safety population included all participants who received at least one dose of INO-4700 or placebo administered by ID injection. Percentage of participants are rounded off to the nearest decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Number analyzed (Participants) | 32 | 33 | 32 | 32 | 31 | 8 | 8 | 8 | 8
percentage of participants | 0 | 6.1 | 3.1 | 0 | 6.5 | 0 | 0 | 12.5 | 0

4. Primary Outcome: Part 1: Geometric Mean Concentration (GMC) of INO-4700 Antigen Specific Binding Antibody at Week 6
Description: Whole blood and serum samples were collected for the cellular immunology assessment. MERS receptor binding domain (RBD) immunoglobulin G (IgG) concentrations in response to administration of INO-4700 in combination with EP were reported as the GMC.
Time Frame: At Week 6
Population: The mITT population included all participants who received at least one dose of the INO-4700 or placebo. 'Overall number of participants analyzed" indicates the number of participants with data available for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: International Units per mL (IU/mL)
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Number analyzed (Participants) | 32 | 31 | 33 | 32 | 31 | 7 | 8 | 8 | 8
International Units per mL (IU/mL) | 4.30 [2.62 to 7.04] | 3.81 [2.38 to 6.11] | 2.29 [1.59 to 3.29] | 3.05 [1.87 to 4.98] | 8.11 [4.37 to 15.04] | 2.37 [1.55 to 3.63] | 4.97 [1.51 to 16.32] | 2.08 [1.06 to 4.08] | 1.75 [0.70 to 4.37]

5. Primary Outcome: Part 1: Geometric Mean Fold Rise (GMFR) of INO-4700 Antigen Specific Binding Antibody at Week 6
Description: Whole blood and serum samples were collected for the cellular immunology assessment. MERS RBD IgG concentrations in response to administration of INO-4700 in combination with EP were reported as the GMFR.
Time Frame: At Week 6
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Number analyzed (Participants) | 32 | 31 | 33 | 32 | 31 | 7 | 8 | 8 | 8
fold rise | 1.93 [1.24 to 3.02] | 2.04 [1.31 to 3.18] | 1.24 [1.01 to 1.52] | 1.40 [1.12 to 1.76] | 3.20 [1.93 to 5.29] | 1.10 [0.94 to 1.28] | 1.09 [0.93 to 1.28] | 1.30 [0.87 to 1.93] | 0.98 [0.92 to 1.06]

6. Primary Outcome: Part 1: Geometric Mean Concentration (GMC) of INO-4700 Antigen Specific Binding Antibody at Week 10
Description: Whole blood and serum samples were collected for the cellular immunology assessment. MERS RBD IgG concentrations in response to administration of INO-4700 in combination with EP were reported as the GMC.
Time Frame: At Week 10
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: International Units per mL (IU/mL)
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Number analyzed (Participants) | 32 | 31 | 33 | 32 | 31 | 7 | 8 | 8 | 8
International Units per mL (IU/mL) | 5.07 [3.09 to 8.32] | 6.68 [3.80 to 11.72] | 3.49 [2.07 to 5.90] | 7.33 [3.56 to 15.09] | 11.92 [6.02 to 23.58] | 1.99 [1.36 to 2.92] | 5.36 [1.88 to 15.25] | 1.84 [0.94 to 3.60] | 1.68 [0.62 to 4.52]

7. Primary Outcome: Part 1: Geometric Mean Fold Rise (GMFR) of INO-4700 Antigen Specific Binding Antibody at Week 10
Description: as for outcome 5
Time Frame: At Week 10
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Number analyzed (Participants) | 32 | 31 | 33 | 32 | 31 | 7 | 8 | 8 | 8
fold rise | 2.31 [1.52 to 3.50] | 3.60 [2.09 to 6.20] | 1.88 [1.24 to 2.84] | 3.38 [1.88 to 6.05] | 4.69 [2.57 to 8.53] | 0.94 [0.84 to 1.05] | 1.22 [0.97 to 1.53] | 1.14 [0.82 to 1.58] | 0.95 [0.76 to 1.19]

8. Primary Outcome: Part 1: Percentage Neutralizing Antibody Responders at Week 6
Description: The immune responses to INO-4700 were measured using assays that included a pseudovirus-based neutralization assay. Immunology blood samples were collected at serial time points. A MERS pseudovirus neutralizing antibody responder was defined as a participant with a sample post-treatment 50% inhibitory dose (ID50) that was >20. Percentage responders were calculated based on number of responders at specified visit divided by number of participants evaluable at specified visit.
Time Frame: At Week 6
Population: as for outcome 4
Measure: Number; unit: percentage of responders
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 31 | 7 | 8 | 8 | 8
percentage of responders | 12.50 | 12.90 | 6.25 | 6.25 | 12.90 | 0 | 0 | 0 | 0

9. Primary Outcome: Part 1: Percentage Neutralizing Antibody Responders at Week 10
Description: as for outcome 8
Time Frame: At Week 10
Population: as for outcome 4
Measure: Number; unit: percentage of responders
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Number analyzed (Participants) | 32 | 30 | 33 | 32 | 31 | 7 | 8 | 8 | 8
percentage of responders | 15.63 | 10.00 | 9.09 | 15.63 | 12.90 | 14.29 | 0 | 0 | 0

10. Primary Outcome: Part 1: Percentage of Antigen Specific Cellular Immune Responders at Week 6
Description: Assessments of cellular immune responses to INO-4700 were performed using the immune response measured by interferon-gamma (IFN-γ) enzyme-linked immunospot (ELISpot) assay on peripheral blood mononuclear cells (PBMCs). A MERS spike ELISpot responder was defined as a participant with a post-treatment level that was > baseline + 2 standard deviations of replicate. Percentage responders were calculated as on number of responders at specified visit divided by number of participants evaluable at specified visit.
Time Frame: At Week 6
Population: as for outcome 4
Measure: Number; unit: percentage of responders
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Number analyzed (Participants) | 28 | 26 | 26 | 27 | 25 | 8 | 8 | 8 | 5
percentage of responders | 14.29 | 11.54 | 0 | 3.70 | 24.00 | 0 | 0 | 0 | 20.00

11. Primary Outcome: Part 1: Percentage of Antigen Specific Cellular Immune Responders at Week 10
Description: as for outcome 10
Time Frame: At Week 10
Population: as for outcome 4
Measure: Number; unit: percentage of responders
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
Number analyzed (Participants) | 31 | 27 | 26 | 29 | 29 | 8 | 8 | 8 | 7
percentage of responders | 6.45 | 7.41 | 23.08 | 24.14 | 17.24 | 0 | 0 | 0 | 14.29

12. Primary Outcome: Part 2: Percentage of Participants With Adverse Events
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have causal relationship with treatment.
Time Frame: From the first dose of the study drug up to the end of the study (up to 68 weeks)
Population: None of the dose groups studied in Part 1 met the immunological criteria for advancement to Part 2. Consequently, the study ended at the conclusion of Part 1 and Part 2 was not conducted.
Arm/Group | Part 2: Parts 2A and 2B
Number analyzed (Participants) | 0

13. Primary Outcome: Part 2: Percentage of Participants With Injection Site Reactions
Description: Reactions arising from the injectable product administration procedure were reported as injection site reactions. Injection site reactions were assessed in accordance with the 'Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials' (FDA Guidance for Industry, September 2007). Local reactions to the injectable product such as pain, tenderness, erythema/redness, and induration/swelling were recorded. Injection site reactions were evaluated starting 30 minutes following the injection.
Time Frame: From the first dose of the study up to the end of the study (up to 68 weeks)
Population: as for outcome 12
Arm/Group | Part 2: Parts 2A and 2B
Number analyzed (Participants) | 0

14. Primary Outcome: Part 2: Percentage of Participants With Adverse Events of Special Interest (AESIs)
Description: An AESI (serious or non-serious) was defined as one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Principal Investigator to the Sponsor can be appropriate. These included respiratory distress syndrome, pneumonia, neurologic, hematologic, immunologic, and other events (including local or systemic SAEs, acute renal failure, SARS-CoV-2 infection, or death). In addition, anxiety and pain related to the EP procedure were monitored.
Time Frame: From Screening up to the end of the study (up to 68 weeks)
Population: as for outcome 12
Arm/Group | Part 2: Parts 2A and 2B
Number analyzed (Participants) | 0

15. Primary Outcome: Part 2: Geometric Mean Concentration (GMC) of INO-4700 Antigen Specific Binding Antibody
Description: Whole blood and serum samples were collected for the cellular immunology assessment. MERS receptor binding domain (RBD) immunoglobulin G (IgG) concentrations in response to administration of INO-4700 in combination were to be assessed.
Time Frame: At Week 12
Population: as for outcome 12
Arm/Group | Part 2: Parts 2A and 2B
Number analyzed (Participants) | 0

16. Primary Outcome: Part 2: Percentage Neutralizing Antibody Responders
Description: The immune responses to INO-4700 were to be measured using assays that included a pseudovirus-based neutralization assay. Immunology blood samples were to be collected at serial timepoints.
Time Frame: At Week 12
Population: as for outcome 12
Arm/Group | Part 2: Parts 2A and 2B
Number analyzed (Participants) | 0

17. Primary Outcome: Part 2: Percentage of Antigen Specific Cellular Immune Responders
Description: Assessments of cellular immune responses to INO-4700 were to be performed using the immune response measured by interferon-gamma (IFN-γ) enzyme-linked immunospot (ELISpot) assay on peripheral blood mononuclear cells (PBMCs).
Time Frame: At Week 12
Population: as for outcome 12
Arm/Group | Part 2: Parts 2A and 2B
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first dose of the study drug up to the end of the study (up to approximately 48.7 weeks)
Description: The safety population included all participants who received at least one dose of INO-4700 or placebo administered by ID injection. None of the dose groups studied in Part 1 met the immunological criteria for advancement to Part 2. Consequently, the study ended at the conclusion of Part 1 and Part 2 was not conducted. Hence, safety data has been reported for Part 1 only.
Arm/Group | Part 1: INO-4700 Group A | Part 1: INO-4700 Group B | Part 1: INO-4700 Group C | Part 1: INO-4700 Group D | Part 1: INO-4700 Group E | Part 1: Placebo Group F | Part 1: Placebo Group G | Part 1: Placebo Group H | Part 1: Placebo Group I
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33 | 0/32 | 0/32 | 0/31 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/33 | 0/32 | 1/32 | 0/31 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/32 | 10/33 | 11/32 | 8/32 | 11/31 | 2/8 | 6/8 | 2/8 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: INO-4700 Group A (N=32) | Part 1: INO-4700 Group B (N=33) | Part 1: INO-4700 Group C (N=32) | Part 1: INO-4700 Group D (N=32) | Part 1: INO-4700 Group E (N=31) | Part 1: Placebo Group F (N=8) | Part 1: Placebo Group G (N=8) | Part 1: Placebo Group H (N=8) | Part 1: Placebo Group I (N=8)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: INO-4700 Group A (N=32) | Part 1: INO-4700 Group B (N=33) | Part 1: INO-4700 Group C (N=32) | Part 1: INO-4700 Group D (N=32) | Part 1: INO-4700 Group E (N=31) | Part 1: Placebo Group F (N=8) | Part 1: Placebo Group G (N=8) | Part 1: Placebo Group H (N=8) | Part 1: Placebo Group I (N=8)
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 3 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 4 | 3 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Red blood cells urine (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 1 | 2 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 4 | 1 | 1 | 2 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT04588428/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT04588428/SAP_001.pdf